CLINICAL TRIAL: NCT03252301
Title: Assessment of Pain in Surgical Patient by PMD 200
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Hospital, Kfar Saba, Israel (Other)
Responsible Party: Principal Investigator, Guy Elad, principal investigator, Meir Hospital, Kfar Saba, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0054-17-MMC
Record Dates: First submitted 2017-08-11; First posted 2017-08-17 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative
Keywords: pain; post operative; surgery; objective
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PMD 200 — finger sensor which estimate objectively the pain level

SUMMARY:
The trial will estimate post-operative pain management in elective surgical patients using the PMD-200 device. The device measures physiological parameters by placing a non-invasive sensor on a fingertip and displays an objective pain level in a 0-100 scale. The pain level will be estimated before surgery (baseline), after surgery and during administration of parenteral analgesia. Treatment and analgesia will be given according to clinical considerations and standard ward protocols. The device measurements won't influence the treatment.

DETAILED DESCRIPTION:
1. Background The key to adequate pain management is assessing its presence, duration and severity, identifying those who require intervention, and evaluating the treatment efficacy. Pain relates to both the noxious input, via peripheral nerves, and to central modulation, thereby, integrating different modalities such as affect, experience or personality. Nociception refers to the peripheral and central nervous system (CNS) processing of information about the internal or external environment, as generated by activation of nociceptors. Typically, noxious stimuli, including tissue injury, activate nociceptors that are present in peripheral structures and that transmit information to the spinal cord dorsal horn (or its trigeminal homologue - the nucleus caudalis). From there, the information continues to the brainstem and ultimately the cerebral cortex, where the perception of pain is generated. The pain is a product of higher brain center processing, whereas nociception can occur in the absence of pain.

   Objective assessment of nociception poses a multitude of challenges. First, sedated or unconscious patients by definition cannot experience pain. Under these circumstances, it is more accurate to assess the nociception level. A body of research suggests that not managing nociception can lead to central changes in pain pathways that predispose individuals to chronic pain states.

   Current "gold-standard" pain assessment tools rely on self-reporting, requiring an individual both to process external information and to communicate this personal experience.

   Circumstances exist where self-reporting is not possible, or where it is unreliable. In these situations, surrogate markers utilize changes in behavioral or physiological parameters. However, their use can be associated with considerable shortcomings. They may be unreliable, hampered by observational bias, or influenced by disease processes or pharmacological interventions. Developing an objective method of pain assessment therefore needs to ensure tools that are sensitive and specific to pain. They need to be observer-independent, not reliant on the patient's ability to communicate and not influenced by disease characteristics.

   A novel measure of nociception is the nociception level (NoL) index. It is based on objective measures related to changes in the autonomic nervous system. The NoL index ranges from 0 to 100 and is based on a nonlinear combination of nociception-related physiologic variables, specifically heart rate, heart rate variability at the 0.15- to 0.4-Hz band power, photoplethysmograph wave amplitude , skin conductance level, number of skin conductance fluctuations, and their time derivatives.

   In the trial the invastigator assume that combination of several parameters into a single one (Nol Index) may have a stronger association with pain intensity than each of the parameters alone.

   Medasense Biometrics Ltd. developed the PMD-200, a nociception/pain monitor that is based on a patented, non-invasive technology enabling objective, continuous assessment of changes in pain level. Information is collected through a finger-mounted probe that monitors changes in multiple pain-related physiological parameters (pulse rate, photoplethismograph amplitude, heart rate variability, skin conductance level and number of skin conductance fluctuations). This information is analyzed using proprietary artificial intelligence algorithms, which convert the physiological data to a real-time nociception Index.

   The rationale for developing the device is to provide caregivers with the ability to measure pain level (or nociception level for unconscious patients) during any procedure and at any time. This information can prevent unnecessary pain, avoid overdose or under usage of analgesic agents, enhance recovery and decrease hospitalization time and costs, while answering the critical need to supervise patients' pain/nociception level.

   The finger probe sensor of PMD-200 collects the following signals:
   1. PhotoPlethysmograph (PPG) - used to optically obtain a volumetric measurement of the finger's tip blood vessels. The trace is generated by light emitted from a LED (~780nm) and collected by a photo diode.
   2. Galvanic Skin Response (GSR) - used to measure the electrical conductance of the skin, which varies with its moisture level. The conductance is obtained by injecting a current between two electrodes placed on the finger and measuring the voltage.
   3. Temperature (TMP) - used to measure the skin temperature using a thermistor.
   4. Accelerometer (ACC) - used to measure finger movements The technology consists of measurements of a number of pain-related physiological parameters that corresponds with the autonomic nervous system's response to pain, and using the company's proprietary algorithms, 'translating' these measurements into an index that represents the pain response, the NoL™ (Nociception Level) Index. This index is displayed on a bedside monitor.

   The measurements taken by the Medasense monitor include galvanic skin response, photoplethysmography , skin temperature and movement .

   All measurements are taken simultaneously using a single finger probe attached to the patient's finger. Miniature sensors are embedded into the probe, which includes reusable and single use components. The finger probe is connected to the bedside monitor for processing of the data.

   Operating the PMD-200 monitor is similar to other standard-of-care systems that track changes in patients' vital functions, such as heart rate, blood pressure or blood oxygen saturation. Such monitors obtain their information from sensing element(s) attached to the patient, display the respective clinical values on a bedside, generate relevant alerts, and maintain records of the information tracked.
2. Methods Population study - electively patients that are going to underwent laparoscopic cholecystectomy.

   1. First measurement will be taken a day before surgery by placing the device on a patient's 3rd finger for 3-5 minutes in a quiet environment. The measurement will be the NOL value (baseline) without pain. The patient will be asked to estimate the pain level using VAS (visual analog scale) score of 0-10.
   2. After determining the NOL value, an IV catheter will be inserted, as required pre-operatively.
   3. The device will continue measuring the pain level while the patient will be asked to estimate the pain level again using VAS .
   4. The patient will be operated.
   5. The patient will receive post-operative analgesia according to ward protocol - PRN IV Dipyrone 1g or PRN IV Paracetamol 1g.
   6. The device will measure pain from 5 minutes before until 20 minutes after analgesics administration. During this time VAS score will be taken. This measure will be taken up to 3 times during the post-operative hospitalization.
   7. The measurement will be taken in a quiet environment without distractions. Any distraction during measurement will be noted as an EVENT.
3. Aims

   1. To examine the response of NoL Index in relation to pain
   2. To develop objective tool to assess the severity of pain in post-operative patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100
* Elective patient for laparoscopic cholecystectomy
* Absence of acute or chronic pain

Exclusion Criteria:

* Pregnancy
* Dementia and mental retardation
* Drugs that influence the autonomic system as beta blocker
* Arrhythmia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
pain level estimation by 1-100 scale by non invasive finger sensor | up to 7 months
  a finger sensor will estimate the pain by a numerical scale of 1-100 in which 1 stand for no pain and 100 stand for severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: haim Paran, MD, Study Chair — clalit

IPD SHARING:
Plan to Share IPD: No